CLINICAL TRIAL: NCT02453516
Title: The Effect of The Serratus Block on Analgesia After Breast Surgery A Randomized Controlled Double-Blinded Study
Brief Title: The Effect of the Serratus Block on Pain Control After Breast Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-0051-E
Record Dates: First submitted 2015-05-13; First posted 2015-05-25 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Anesthesia
Keywords: Serratus Block; Breast Surgery
MeSH Terms: interventions — Ropivacaine; Epinephrine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Serratus Block Group (Experimental): Patients will receive a preoperative ultrasound-guided serratus block with 0.4ml/kg (max.30ml) of ropivacaine 0.5% with 1:4000,000 epinephrine injected between the serratus anterior (superficial) and external intercostal (deep) muscles followed by subsequent general anesthesia
  Interventions: Procedure: Serratus Block; Drug: ropivacaine; Drug: epinephrine
- Placebo Block - Control Group (Placebo Comparator): Patients will receive a preoperative placebo injection with a subcutaneous injection of 1ml normal sterile saline solution in the midaxillary line and the ultrasound probe will be used to simulate the pressure and block duration associated with the serratus block. These patients will then receive general anesthesia.
  Interventions: Procedure: Placebo Block; Other: sterile saline

INTERVENTIONS:
Procedure: Serratus Block — Ultrasound-guided nerve block using ropivacaine 0.5% (0.4ml/kg) injected between the serratus anterior and external intercostal muscles
  Arms: Serratus Block Group
Procedure: Placebo Block — Subcutaneous injection of 1ml sterile normal saline solution in the midaxillary line
  Other Names: Control Group - Placebo Comparator
  Arms: Placebo Block - Control Group
Drug: ropivacaine — Drug indicated for regional anesthesia
  Other Names: Naropin HCL
  Arms: Serratus Block Group
Drug: epinephrine — Drug indicated to prolong the action of regional anesthesia
  Other Names: Adrenaline Chloride
  Arms: Serratus Block Group
Other: sterile saline — Neutral injection (no drug involved)
  Other Names: Sodium Chloride
  Arms: Placebo Block - Control Group

SUMMARY:
Surgery for breast cancer is associated with significant pain. The serratus nerve block targets the interfascial plane either below or above the serratus muscle, blocking thereby the lateral cutaneous branches of the intercostal nerves. The purpose of this randomized controlled double-blinded study is to see whether the addition of a serratus nerve block to a general anesthesia results in a better postoperative pain control in patients undergoing surgery for breast cancer.

DETAILED DESCRIPTION:
The prevalence of severe acute postoperative pain after breast surgery is high. Regional anesthesia has the potential to provide superior pain relief with fewer side effects compared to standard systemic opioid therapy. The search for a regional anesthesia technique for breast surgery has been ongoing as this technique needs to be time efficient, relatively risk-free and also practicable in an out-patient setting. The serratus block is a promising technique that may combine these advantages.

ELIGIBILITY:
Inclusion Criteria:

* ASA I to III (American Society of Anesthesiologists Physical Status Classification System)
* undergoing unilateral primary or secondary breast surgery for cancer, specifically: lumpectomies with sentinel node biopsy or partial mastectomies or simple mastectomies, with or without sentinel node biopsy
* day surgery procedures

Exclusion Criteria:

* inability to understand or to provide consent
* inability or unwillingness to comply with required follow-up assessments
* psychiatric disorder affecting patient assessment
* contraindication to regional anesthesia, e.g., coagulopathy
* allergy to local anesthestic
* chronic pain and/or chronic use of opioids with a daily use of over 30mg oxycodone or equivalent per day
* contraindication to a component of multimodal analgesia
* preexisting neuropathy with motor or sensory deficits in the area of the anterolateral chest wall
* infection near the injection site
* pregnancy
* BMI >35
* complication or adverse events unrelated to the study intervention that precludes evaluation of the primary and secondary outcomes

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10-29 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Post-operative pain scores | Scores collected @ 3 different time points: admission to phase I recovery (PACU), admission to phase II recovery (day surgery unit), and discharge from day surgery unit The total time time is estimated to be up to 6 hours..
  The patient's level of pain in the postoperative period will be evaluated by the use of a 100mm Visual Analogue Scale (VAS). The mean of these scores at the 3 different time points will be calculated.

SECONDARY OUTCOMES:
Intraoperative opioid consumption | Duration of actual surgical procedure
Post-operative opioid consumption | End of surgical procedure until 7 days after surgery
Duration phase I and phase II recovery | Admission to phase I recovery (PACU) until discharge from phase II recovery, total time is estimated up to 6 hours,
  Duration of stay in PACU and in surgical day care
Opioid side-effects | End of surgical procedure to 7 days following surgery
  Opioid-related side effects (nausea, vomiting, pruritis)
Block-related side-effects | Completion of block to 3 months postoperatively
  Presence/absence of block-related side effects such as bruising, infection, systemic toxicity, persistent numbness or shoulder weakness
Satisfaction with analgesia | End of surgical procedure to 3 months postoperatively
  Scale of 0-10 (0=Not Satisfied, 10=Very Satisfied)
Quality of recovery score (QoR) | Discharge from hospital until 24 hours post-op
  Completion of questionnaire (QoR) done by patient.
Pain assessment | Assessment to be done again @ 6 weeks and 3 months postoperatively. Simple question requiring a yes or no response.
  Persistent postsurgical pain

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brull, MD FRCP, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Abdallah FW, Patel V, Madjdpour C, Cil T, Brull R. Quality of recovery scores in deep serratus anterior plane block vs. sham block in ambulatory breast cancer surgery: a randomised controlled trial. Anaesthesia. 2021 Sep;76(9):1190-1197. doi: 10.1111/anae.15373. Epub 2021 Jan 25. PMID 33492696